CLINICAL TRIAL: NCT03124836
Title: Accuracy of Methemoglobin Measurement of Various Rainbow Pulse Oximeter Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR19427-BICK0001
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- R2-25 Sensor (Experimental): All subjects will be enrolled in the test group and will receive R2-25 Pulse Oximeter Sensor
  Interventions: Device: Pulse Oximeter Sensor

INTERVENTIONS:
Device: Pulse Oximeter Sensor

SUMMARY:
In this study, the level of methemoglobin (HbMet) will be increased in a controlled manner by administering sodium nitrite intravenously in healthy volunteers. The accuracy of the noninvasive HbMet measurement by a Pulse Oximeter Sensor will be assessed by comparison to blood measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female, aged ≥18 and <50.
2. The subject is in good general health with no evidence of any medical problems.
3. The subject is fluent in both written and spoken English.
4. The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

1. The subject is obese (BMI>30).
2. The subject has a known history of heart disease, lung disease, kidney or liver disease.
3. Diagnosis of asthma, sleep apnea, or use of CPAP.
4. Subject has diabetes.
5. Subject has a clotting disorder.
6. The subject has a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
7. The subject has any other serious systemic illness.
8. The subject is a current smoker.
9. Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
10. The subject has a history of fainting or vasovagal response.
11. The subject has a history of sensitivity to local anesthesia or allergy to the study drugs.
12. The subject has a diagnosis of Raynaud's disease.
13. The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
14. The subject is pregnant, lactating or trying to get pregnant.
15. The subject has a history of migraine headaches.
16. Th subject is currently taking antidepressants.
17. The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
18. The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2009-12-17 (Actual); Study Completion 2009-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- R2-25 Sensor: All subjects will be enrolled in the test group and will receive R2-25 Pulse Oximeter Sensor
  Pulse Oximeter Sensor
Period: Overall Study
Arm/Group | R2-25 Sensor
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | R2-25 Sensor
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Methemoglobin Measurement by Arms Calculation
Description: Accuracy willl be determined by comparing the noninvasive blood methemoglobin measurement (expressed as a percentage of total hemoglobin) of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square(Arms) error value.In order to obtain the Arms value, the blood sample methemoglobin value is subtracted from the pulse oximeter methemoglobin value for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours
Measure: Number; unit: percentage of total hemoglobin
Arm/Group | R2-25 Sensor
Number analyzed (Participants) | 28
percentage of total hemoglobin | 0.48

ADVERSE EVENTS:
Arm/Group | R2-25 Sensor
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less